CLINICAL TRIAL: NCT05795829
Title: First in Man Study to Evaluate the Safety and Efficacy of Disposable Intravascular Ultrasound Ablation Catheters and Ultrasound Ablation Instrument in the Treatment of Essential Hypertension
Brief Title: Ultrasound Ablation for Essential Hypertension（FIM）
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPCTP-2021-004
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Uncontrolled Essential Hypertension
Keywords: Ultrasound Ablation Catheter; Renal Sympathetic Denervation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disposable Intravascular Ultrasound Ablation Catheter and Ultrasound Ablation Instrument (Experimental): All subjects will receive treatment from the disposable intravascular ultrasound ablation catheter.
  Interventions: Device: disposable intravascular ultrasound ablation catheter and ultrasound ablation instrument

INTERVENTIONS:
Device: disposable intravascular ultrasound ablation catheter and ultrasound ablation instrument — Disposable intravascular ultrasound ablation catheters (used with an ultrasound ablation instrument) can use ultrasound energy to block sympathetic activity in the renal arteries.

SUMMARY:
To evaluate the safety and feasibility of disposable intravascular ultrasound ablation catheter and ultrasound ablation instrument in the treatment of essential hypertension.

DETAILED DESCRIPTION:
Feasibility Research This is a prospective, small-sample, single-group study. A total of 10 subjects are planned to be included in this study. Disposable intravascular catheter and instrument are used for intravascular ultrasound ablation. All participants will be followed up by telephone or outpatient at 1, 2 and 6 months post-procedure, with procedural success rate as the primary endpoint. At the same time, the incidence of adverse events will be observed to make a preliminary evaluation of the safety and feasibility of disposable intravascular catheter and instrument, and to provide data support for the second-stage confirmatory study.

In feasibility research, statistical analysis of data will be performed after 30 days postoperative follow-up of the subjects, and the safety and feasibility of disposable intravascular catheter and instrument will be preliminarily evaluated before entering the stage of confirmatory trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 and≤80 years old, no gender limitation;
2. Two or more antihypertensive drugs should be statically taken for at least 4 weeks before randomization and the prescribed dose should be ≥ 50% of the manufacturer's maximum dose， angiotensin-converting enzyme inhibitor (ACEI) (or angiotensin-Ⅱ receptor antagonist (ARB)) and calcium channel blocker (CCB) (or thiazide diuretic) are required to be used in combination. Blood pressure meets the following conditions: 1) office systolic blood pressure (SBP)≥150mmHg and<180mmHg; 2) office diastolic blood pressure (DBP) ≥90mmHg;
3. 24-hour ambulatory systolic blood pressure: ≥135 mmHg and <170 mmHg;
4. A recorded history of essential hypertension;
5. Understands the purpose of this study, and is willing to sign the Informed Consent and complete clinical follow-up.

Exclusion Criteria:

1. Ineligible renal artery anatomy including : (1) multiple renal arteries, (2) main renal artery diameter <4mm or length <20mm, (3) renal artery stenosis > 50% in the main renal artery, (4) atherosclerosis of the renal artery, renal artery aneurysm, fibromuscular dysplasia or calcification, (5) pre-existing renal stent, (6) single kidney
2. Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2
3. Type Ⅰ diabetes mellitus or poorly controlled type Ⅱ diabetes mellitus (defined as plasma Hb1Ac≥ 9.0% or 24-hour urinary protein quantification >1g/24h or proliferative retinopathy)
4. Postural hypotension
5. Recent vascular events: Experienced acute myocardial infarction, unstable angina, syncope, or cerebrovascular accident within 3 months of the screening period
6. Possible secondary hypertension
7. Respiratory support: The individual requires long-term oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea
8. Life expectancy <1 year
9. Female who is pregnant, nursing, or planning to become pregnant
10. Subjects who are currently enrolled in another clinical trial and have not completed their primary endpoint
11. Subjects who are allergic to contrast medium
12. Subjects who are unsuitable for the trial ，because of poor patient compliance or other reasons judged by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Procedural success | Before discharge (post-procedure), up to 7 days
  Procedural success was defined as the absence of renal arterial related complication during the subject's hospitalization based on the device success.

SECONDARY OUTCOMES:
Change in average 24-hour/night-time ambulatory Systolic Blood Pressure (SBP) | 1 month, 2months, 6 months post-procedure
Change in average 24-hour/daytime/night-time ambulatory Diastolic Blood Pressure (DBP) | 1 month, 2months, 6 months post-procedure
Change in average daytime ambulatory Systolic Blood Pressure (SBP) | 1 month, 2months, 6 months post-procedure
Change in office systolic blood pressure | 1 month, 2 months, 6 months post-procedure
Change in office diastolic blood pressure | 1 month, 2 months, 6 months post-procedure
Device success | immediate post-procedure
Incidence of achieving target office systolic blood pressure | 1 month, 2 months, 6 months post-procedure
Significant embolic events resulting in end-organ damage | 1 month, 2 months, 6 months post-procedure
Incidence of acute myocardial infarction, stroke, transient ischemic attack, cerebrovascular accident | 1 month, 2 months, 6 months post-procedure
End-stage renal disease | 1 month, 2 months, 6 months post-procedure
Renal artery or vascular complications requiring intervention | 1 month, 2 months, 6 months post-procedure
Significant (50%) and severe (75%) new onset renal stenosis | 6 months post-procedure
Severe access site complications | 1 month, 2 months, 6 months post-procedure
Incidence of adverse events | 1 month, 2 months, 6 months post-procedure
Stability of ultrasonic ablation instrument | immediate post-procedure
  Whether the instrument has failed during the use of the device, and whether the fault can be recovered.
Interface friendliness of ultrasonic ablation instrument | immediate post-procedure
  It is defined as whether the operation interface and difficulty of operation of the instrument are convenient.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, Study Chair — The Second Affiliated Hospital of Harbin Medical University; Jing Huang, Study Chair — The Second Affiuated Hospital of Chongqing Medical University
Locations (2):
- China (2):
  - The Second Affiuated Hospital of Chongqing Medical University, Chongqing
  - The Second Affiliated Hospital of Harbin Medical University, Harbin